CLINICAL TRIAL: NCT02053012
Title: Investigating Reaction Time Among Children Who Snore
Status: Completed | Type: Observational
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00003
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PVT-192
  Interventions: Device: PVT-192

INTERVENTIONS:
Device: PVT-192 — PVT-192 Psychomotor Vigilance Task Monitor is a hand-held, self-contained system used for repetitive reaction time measurement.

SUMMARY:
The investigators feel that children who have OSA or sleep-disordered breathing may have a different reaction time than normal variants. Children who have OSA are known to have behavioral and sleep patterns that are different. It makes sense their reaction time may be different than normal as well. We plan to measure reaction times via a 10 minute psychomotor vigilance test device in children who snore who are coming in for a sleep study or for adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand how to perform reaction time test and complete without assistance.

Exclusion Criteria:

* Children who are unable to understand or perform test or parents refusal.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who snore and are coming to Nationwide Children's for a sleep study or adenotonsillectomy.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-01; Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Reaction time | 10 minutes
  We plan to measure reaction times via a 10 minute psychomotor vigilance test (PVT, Ambulatory Monitoring Inc., NY) device.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States